CLINICAL TRIAL: NCT03236064
Title: Conversion of Seddon III Nerve Injury to Seddon I/II Nerve Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: WellSpan Health (Other)
Collaborators: Neuraptive Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 696230-1
Record Dates: First submitted 2016-07-25; First posted 2017-08-01 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Injury of Other Nerves at Wrist and Hand Level of Unspecified Arm, Initial Encounter
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nerve injury to palm and fingers (Experimental): Adult patients with acute clean nerve transections of the higher arm injuries in the forearm, wrist, palm and digits of the hand will be recruited
  Interventions: Drug: Polyethylene Glycols

INTERVENTIONS:
Drug: Polyethylene Glycols — Demonstrate more rapid and increased return of function by PEG-fusion compared to best current nerve repair techniques

SUMMARY:
This study will evaluate the safety and efficacy of PEG 3350 for use in nerve repair.

DETAILED DESCRIPTION:
To demonstrate more rapid and increased return of function by PEG-fusion compared to the best current nerve repair techniques. Neurorrhaphy is not new, being performed now for over 150 years much research has been performed. PEG-Axon fusion on the other hand is relatively new in mammals. Success has already been obtained by two institutions in the rat sciatic nerve transections, demonstrating rapid return of behavioral function4. These however are very controlled injuries and unclear how well these will translate into human studies. For this reason 3 separate clinical studies in increasing order of complexity are proposed.

The first study proposed will be PEG fusion in digital nerve lacerations. Two goals will be demonstrated; improved innervation density and improved innervation threshold compared to traditional repair, and complication rate similar or less than traditional repair. This will demonstrate the safety and efficacy of the procedure.

ELIGIBILITY:
* Isolated nerve transections of the digits, forearm, wrist, and palm will be included.
* Class III nerve injury (Sunderland's 4th or 5th degree injury)
* Nerve injuries that can be prepared using minimal or acceptable tension (according to surgeon discretion).
* Pregnant and breastfeeding women cannot participate because of possible unknown and unpredictable risks to the unborn child.
* Injuries beyond 24 hours will be excluded

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-05; Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
To demonstrate more rapid and increased return of function by PEG-fusion compared to the best current nerve repair techniques | 12 months
  Three goals will be demonstrated; improved innervation density and improved innervation threshold compared to traditional repair, rapid return of motor function and complication rate similar or less than traditional repair. This will demonstrate the safety and efficacy of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Trevino, MD, Principal Investigator — WellSpan York Hospital
Locations (1):
- WellSpanYork Hospital, York, Pennsylvania, United States